CLINICAL TRIAL: NCT05823935
Title: Laparoscopic Versus Vaginal Cuff Closure During Laparoscopic Hysterectomy in Benign Gynecological Lesions
Brief Title: Laparoscopic Versus Vaginal Cuff Closure During LH in Benign Gynecological Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD.22.10.703
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Uterine Diseases
Keywords: TLH; Bakay purse string
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bakay purse string group (Active Comparator): Bakay purse string will be used to close the vaginal cuff after total laparoscopic hysterectomy for benign lesions.
  Interventions: Procedure: Bakay purse string
- Cuff closure via vaginal route group (Active Comparator): Vaginal cuff closure via vaginal route with continuous locked suturing will be used to close the vaginal cuff after total laparoscopic hysterectomy for benign lesions.
  Interventions: Procedure: Cuff closure via vaginal route group

INTERVENTIONS:
Procedure: Bakay purse string — After developing the bladder flap, Vicryl polyglactin 910 sutures (Ethicon, Inc, Somerville, NJ) will be placed on the line between the cervicovaginal junction and the bladder starting at either 4 to 3 o'clock or 8 to 9 o'clock, as anchor sutures. Paying attention not to get closer than 1 cm to the bladder, the first suture will be passed from 4 o'clock to 3 o'clock and continued circumferentially in a full-thickness purse string fashion through 3, 1, 10, 8, 7, 5 o'clock completing a circle while including both uterosacral ligaments.
  Arms: Bakay purse string group
Procedure: Cuff closure via vaginal route group — After the uterus will be removed via vaginal route, vaginal cuff ends will be grasped via vaginal approach and sutured continuous locked sutures using Vicryl polyglactin 910 sutures in one layer.
  Arms: Cuff closure via vaginal route group

SUMMARY:
To compare vaginal cuff closure via Bakay purse string with vaginal cuff closure via vaginal route with continuous locked suturing after total laparoscopic hysterectomy for benign lesions.

DETAILED DESCRIPTION:
The objective of the present study is to compare 2 different methods for vaginal cuff closure after total laparoscopic hysterectomy for benign lesions regarding operative time, vaginal length, vaginal cuff dehiscene, hematoma formation. The first method is the Bakay purse string and the second is the closure of the vault via vaginal route with continuous locked suturing.

ELIGIBILITY:
Inclusion Criteria:

* Benign uterine lesions e.g fibroid, adenomyosis,…etc.
* Patient acceptance to undergo laparoscopic hysterectomy.

Exclusion Criteria:

* Gynecological malignancy.
* Low corporeal myoma obsecuring cervicovaginal junction.
* History of extensive abdominal surgery other than cesarean section.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Total operative time | From start to end of operation
  The time between placement of the operative ports and successful closure of the vaginal cuff
Operative time for colpotomy and vaginal cuff closure | From start colpotomy to end of vaginal cuff closure
  The time between first anchor suture placement and successful closure of the vaginal cuff

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Elashry, MSc, Principal Investigator — Mansoura University; Hamed M Youssef, MD, Study Chair — Mansoura University; Maged R Elshamy, MD, Study Director — Mansoura University; Mahmoud M Awad, MD, Study Director — Mansoura University; Mohamed S Abdelhafez, MD, Study Director — Mansoura University
Locations (1):
- Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt